CLINICAL TRIAL: NCT01269697
Title: Lutein Influence on Macula of Persons Issued From Amd Parents
Acronym: LIMPIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHUBX 2009/31
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Persons Issued From Amd Parents
Keywords: AMD; food supplementation; macular pigments; luthéine; zéaxanthine; visual acuity; prevention; genetique risk

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutrof (Active Comparator): patient receive the treatment of Nutrof Total
  Interventions: Dietary Supplement: Nutrof Total
- Placebo of Nutrof (Placebo Comparator): Patient receive the treatment of the placebo of Nutrof Total
  Interventions: Dietary Supplement: Placebo Nutrof total

INTERVENTIONS:
Dietary Supplement: Nutrof Total — 2 capsules 2 times per day during 6 month
  Arms: Nutrof
Dietary Supplement: Placebo Nutrof total — 2 capsules 2 times per day during 6 month
  Arms: Placebo of Nutrof

SUMMARY:
Age-related macular degeneration (AMD) is a degenerative disease of the centre of the retina (named macula) and is the leading cause of blindness in industrialized countries. There is growing interest in the potential preventive role of two carotenoids (lutein and zeaxanthin) of dietary origin, which specifically accumulate in the macula, where they form the macular pigment. A first step towards the demonstration of a preventive effect of macular pigment for AMD consists in the evaluation of the effect of lutein and zeaxanthin supplementation on their plasma and retinal concentrations.

DETAILED DESCRIPTION:
The objective of this study is to estimate the efficiency of a nutritonal supplementation with lutein and zeaxanthin to increase their plasma concentration and the density of macular pigment, in subjects at high genetic risk for AMD (1st generation stemming from parent affected by DMLA). This study is a multicentric, double blind, randomized clinical trial of supplementation versus placebo

ELIGIBILITY:
Inclusion Criteria:

* Men or women 40 to 70 years old
* Presenting histories of wet AMD with their father or their mother or 2
* Visual acuity of 20/25 or better (ETDRS)
* The presence of a AMD in one eye is possible
* Enlightened consent writes, dated and signed by the participant and the investigator above all examination required by the research.
* Subject agreeing to be registered in the national file
* Affiliated or profitable subject of a national insurance scheme

Exclusion Criteria:

* Presence of signs of AMD in both eyes (if AMD in one eye, inclusion for the other eye is possible)
* Histories of the other evolutionary eye pathologies susceptible to complicate the evaluation of the AMD and of the visual acuity (severe glaucoma, strong nearsightedness (superior or more equal in - 6 dioptres), the other severe rétinopathie)
* Subject with history of cataract surgery
* Opaqueness preventing the evaluation of the photos of the retina (cataract, corneal dystrophy)
* Supplementation with food complements in the year which precedes (cf. appendix 2 of the protocol)
* Participation in another clinical trial during 30 days which precede
* Subjects not compliants
* Subjects not flatware by the system of social security
* Subjects under guardianship judicial

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The main assessment criterion is the measure of the evolution of the density of the macular pigment after 6 months of supplementation | 6 months after stop of the supplementation
  Difference in measures of the density of the macular pigment at baseline and 6 months after stop of the supplementation

SECONDARY OUTCOMES:
Measure of the modification of the visual acuteness with correction | 12 months
Measure of the cognitive capacities | 12 months
Measure rates plasmatiques of fatty acids | 12 months
Measure of the evolution of the density of the macular pigment during supplementation and after stop of the supplementation | 1 year
  Measure of the density of the macular pigment before supplementation, in 3 and 6 months during the supplementation and in 3 and 6 months after stop of the supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François KOROBELNIK, Professor, Principal Investigator — University Hospital Bordeaux, France; Geneviève CHENE, Professor, Study Chair — University Hospital Bordeaux, France
Locations (2):
- France (2):
  - Unité Médicale Rétine Neuro-Ophtalmologie - Service d'Ophtalmologie - Hopital Pellegrin, Bordeaux
  - Service Ophtalmologie - Hôpital général CHU de Dijon, Dijon

REFERENCES:
- [Background] Resnikoff S, Pascolini D, Etya'ale D, Kocur I, Pararajasegaram R, Pokharel GP, Mariotti SP. Global data on visual impairment in the year 2002. Bull World Health Organ. 2004 Nov;82(11):844-51. Epub 2004 Dec 14. PMID 15640920
- [Background] Jager RD, Mieler WF, Miller JW. Age-related macular degeneration. N Engl J Med. 2008 Jun 12;358(24):2606-17. doi: 10.1056/NEJMra0801537. No abstract available. PMID 18550876
- [Background] Age-Related Eye Disease Study Research Group. A randomized, placebo-controlled, clinical trial of high-dose supplementation with vitamins C and E, beta carotene, and zinc for age-related macular degeneration and vision loss: AREDS report no. 8. Arch Ophthalmol. 2001 Oct;119(10):1417-36. doi: 10.1001/archopht.119.10.1417. PMID 11594942
- [Background] Whitehead AJ, Mares JA, Danis RP. Macular pigment: a review of current knowledge. Arch Ophthalmol. 2006 Jul;124(7):1038-45. doi: 10.1001/archopht.124.7.1038. PMID 16832030
- [Background] Antioxidant status and neovascular age-related macular degeneration. Eye Disease Case-Control Study Group. Arch Ophthalmol. 1993 Jan;111(1):104-9. doi: 10.1001/archopht.1993.01090010108035. PMID 7678730
- [Background] Gale CR, Hall NF, Phillips DI, Martyn CN. Lutein and zeaxanthin status and risk of age-related macular degeneration. Invest Ophthalmol Vis Sci. 2003 Jun;44(6):2461-5. doi: 10.1167/iovs.02-0929. PMID 12766044
- [Background] Delcourt C, Carriere I, Delage M, Barberger-Gateau P, Schalch W; POLA Study Group. Plasma lutein and zeaxanthin and other carotenoids as modifiable risk factors for age-related maculopathy and cataract: the POLA Study. Invest Ophthalmol Vis Sci. 2006 Jun;47(6):2329-35. doi: 10.1167/iovs.05-1235. PMID 16723441
- [Background] Tan JS, Wang JJ, Flood V, Rochtchina E, Smith W, Mitchell P. Dietary antioxidants and the long-term incidence of age-related macular degeneration: the Blue Mountains Eye Study. Ophthalmology. 2008 Feb;115(2):334-41. doi: 10.1016/j.ophtha.2007.03.083. Epub 2007 Jul 30. PMID 17664009
- [Background] Cho E, Hankinson SE, Rosner B, Willett WC, Colditz GA. Prospective study of lutein/zeaxanthin intake and risk of age-related macular degeneration. Am J Clin Nutr. 2008 Jun;87(6):1837-43. doi: 10.1093/ajcn/87.6.1837. PMID 18541575
- [Background] VandenLangenberg GM, Mares-Perlman JA, Klein R, Klein BE, Brady WE, Palta M. Associations between antioxidant and zinc intake and the 5-year incidence of early age-related maculopathy in the Beaver Dam Eye Study. Am J Epidemiol. 1998 Jul 15;148(2):204-14. doi: 10.1093/oxfordjournals.aje.a009625. PMID 9676703
- [Background] Cho E, Seddon JM, Rosner B, Willett WC, Hankinson SE. Prospective study of intake of fruits, vegetables, vitamins, and carotenoids and risk of age-related maculopathy. Arch Ophthalmol. 2004 Jun;122(6):883-92. doi: 10.1001/archopht.122.6.883. PMID 15197064
- [Background] van Leeuwen R, Boekhoorn S, Vingerling JR, Witteman JC, Klaver CC, Hofman A, de Jong PT. Dietary intake of antioxidants and risk of age-related macular degeneration. JAMA. 2005 Dec 28;294(24):3101-7. doi: 10.1001/jama.294.24.3101. PMID 16380590
- [Background] Beatty S, Murray IJ, Henson DB, Carden D, Koh H, Boulton ME. Macular pigment and risk for age-related macular degeneration in subjects from a Northern European population. Invest Ophthalmol Vis Sci. 2001 Feb;42(2):439-46. PMID 11157880
- [Background] Bone RA, Landrum JT, Mayne ST, Gomez CM, Tibor SE, Twaroska EE. Macular pigment in donor eyes with and without AMD: a case-control study. Invest Ophthalmol Vis Sci. 2001 Jan;42(1):235-40. PMID 11133874
- [Background] Bernstein PS, Zhao DY, Wintch SW, Ermakov IV, McClane RW, Gellermann W. Resonance Raman measurement of macular carotenoids in normal subjects and in age-related macular degeneration patients. Ophthalmology. 2002 Oct;109(10):1780-7. doi: 10.1016/s0161-6420(02)01173-9. PMID 12359594
- [Background] Obana A, Hiramitsu T, Gohto Y, Ohira A, Mizuno S, Hirano T, Bernstein PS, Fujii H, Iseki K, Tanito M, Hotta Y. Macular carotenoid levels of normal subjects and age-related maculopathy patients in a Japanese population. Ophthalmology. 2008 Jan;115(1):147-57. doi: 10.1016/j.ophtha.2007.02.028. PMID 18166409
- [Background] Hammond BR Jr, Johnson EJ, Russell RM, Krinsky NI, Yeum KJ, Edwards RB, Snodderly DM. Dietary modification of human macular pigment density. Invest Ophthalmol Vis Sci. 1997 Aug;38(9):1795-801. PMID 9286268
- [Background] Berendschot TT, Goldbohm RA, Klopping WA, van de Kraats J, van Norel J, van Norren D. Influence of lutein supplementation on macular pigment, assessed with two objective techniques. Invest Ophthalmol Vis Sci. 2000 Oct;41(11):3322-6. PMID 11006220
- [Background] Bone RA, Landrum JT, Guerra LH, Ruiz CA. Lutein and zeaxanthin dietary supplements raise macular pigment density and serum concentrations of these carotenoids in humans. J Nutr. 2003 Apr;133(4):992-8. doi: 10.1093/jn/133.4.992. PMID 12672909
- [Background] Koh HH, Murray IJ, Nolan D, Carden D, Feather J, Beatty S. Plasma and macular responses to lutein supplement in subjects with and without age-related maculopathy: a pilot study. Exp Eye Res. 2004 Jul;79(1):21-7. doi: 10.1016/j.exer.2004.03.001. PMID 15183097
- [Background] Wenzel AJ, Gerweck C, Barbato D, Nicolosi RJ, Handelman GJ, Curran-Celentano J. A 12-wk egg intervention increases serum zeaxanthin and macular pigment optical density in women. J Nutr. 2006 Oct;136(10):2568-73. doi: 10.1093/jn/136.10.2568. PMID 16988128
- [Background] Bone RA, Landrum JT, Cao Y, Howard AN, Alvarez-Calderon F. Macular pigment response to a supplement containing meso-zeaxanthin, lutein and zeaxanthin. Nutr Metab (Lond). 2007 May 11;4:12. doi: 10.1186/1743-7075-4-12. PMID 17498306
- [Background] Thurnham DI, Tremel A, Howard AN. A supplementation study in human subjects with a combination of meso-zeaxanthin, (3R,3'R)-zeaxanthin and (3R,3'R,6'R)-lutein. Br J Nutr. 2008 Dec;100(6):1307-14. doi: 10.1017/S0007114508971336. Epub 2008 Apr 11. PMID 18405400
- [Background] Huang LL, Coleman HR, Kim J, de Monasterio F, Wong WT, Schleicher RL, Ferris FL 3rd, Chew EY. Oral supplementation of lutein/zeaxanthin and omega-3 long chain polyunsaturated fatty acids in persons aged 60 years or older, with or without AMD. Invest Ophthalmol Vis Sci. 2008 Sep;49(9):3864-9. doi: 10.1167/iovs.07-1420. Epub 2008 Apr 30. PMID 18450596
- [Background] Schalch W, Cohn W, Barker FM, Kopcke W, Mellerio J, Bird AC, Robson AG, Fitzke FF, van Kuijk FJ. Xanthophyll accumulation in the human retina during supplementation with lutein or zeaxanthin - the LUXEA (LUtein Xanthophyll Eye Accumulation) study. Arch Biochem Biophys. 2007 Feb 15;458(2):128-35. doi: 10.1016/j.abb.2006.09.032. Epub 2006 Nov 7. PMID 17084803
- [Background] Trieschmann M, Beatty S, Nolan JM, Hense HW, Heimes B, Austermann U, Fobker M, Pauleikhoff D. Changes in macular pigment optical density and serum concentrations of its constituent carotenoids following supplemental lutein and zeaxanthin: the LUNA study. Exp Eye Res. 2007 Apr;84(4):718-28. doi: 10.1016/j.exer.2006.12.010. Epub 2006 Dec 19. PMID 17306793
- [Background] Johnson EJ, Chung HY, Caldarella SM, Snodderly DM. The influence of supplemental lutein and docosahexaenoic acid on serum, lipoproteins, and macular pigmentation. Am J Clin Nutr. 2008 May;87(5):1521-9. doi: 10.1093/ajcn/87.5.1521. PMID 18469279
- [Background] De Jong PT, Klaver CC, Wolfs RC, Assink JJ, Hofman A. Familial aggregation of age-related maculopathy. Am J Ophthalmol. 1997 Dec;124(6):862-3. doi: 10.1016/s0002-9394(14)71715-5. No abstract available. PMID 9402844
- [Background] Klaver CC, Wolfs RC, Assink JJ, van Duijn CM, Hofman A, de Jong PT. Genetic risk of age-related maculopathy. Population-based familial aggregation study. Arch Ophthalmol. 1998 Dec;116(12):1646-51. doi: 10.1001/archopht.116.12.1646. PMID 9869796
- [Background] Young TL. Molecular genetics of human myopia: an update. Optom Vis Sci. 2009 Jan;86(1):E8-E22. doi: 10.1097/OPX.0b013e3181940655. PMID 19104467
- [Background] Nolan JM, Stack J, O' Donovan O, Loane E, Beatty S. Risk factors for age-related maculopathy are associated with a relative lack of macular pigment. Exp Eye Res. 2007 Jan;84(1):61-74. doi: 10.1016/j.exer.2006.08.016. Epub 2006 Nov 1. PMID 17083932
- [Background] Nolan JM, Stack J, O'connell E, Beatty S. The relationships between macular pigment optical density and its constituent carotenoids in diet and serum. Invest Ophthalmol Vis Sci. 2007 Feb;48(2):571-82. doi: 10.1167/iovs.06-0864. PMID 17251452
- [Background] Zeimer M, Hense HW, Heimes B, Austermann U, Fobker M, Pauleikhoff D. [The macular pigment: short- and intermediate-term changes of macular pigment optical density following supplementation with lutein and zeaxanthin and co-antioxidants. The LUNA Study]. Ophthalmologe. 2009 Jan;106(1):29-36. doi: 10.1007/s00347-008-1773-4. German. PMID 18551295
- [Background] Akbaraly NT, Faure H, Gourlet V, Favier A, Berr C. Plasma carotenoid levels and cognitive performance in an elderly population: results of the EVA Study. J Gerontol A Biol Sci Med Sci. 2007 Mar;62(3):308-16. doi: 10.1093/gerona/62.3.308. PMID 17389729
- [Background] Cunnane SC, Plourde M, Pifferi F, Begin M, Feart C, Barberger-Gateau P. Fish, docosahexaenoic acid and Alzheimer's disease. Prog Lipid Res. 2009 Sep;48(5):239-56. doi: 10.1016/j.plipres.2009.04.001. Epub 2009 Apr 10. PMID 19362576
- [Background] Rinaldi P, Polidori MC, Metastasio A, Mariani E, Mattioli P, Cherubini A, Catani M, Cecchetti R, Senin U, Mecocci P. Plasma antioxidants are similarly depleted in mild cognitive impairment and in Alzheimer's disease. Neurobiol Aging. 2003 Nov;24(7):915-9. doi: 10.1016/s0197-4580(03)00031-9. PMID 12928050
- [Background] Johnson EJ, McDonald K, Caldarella SM, Chung HY, Troen AM, Snodderly DM. Cognitive findings of an exploratory trial of docosahexaenoic acid and lutein supplementation in older women. Nutr Neurosci. 2008 Apr;11(2):75-83. doi: 10.1179/147683008X301450. PMID 18510807
- [Background] Wolf-Schnurrbusch UE, Roosli N, Weyermann E, Heldner MR, Hohne K, Wolf S. Ethnic differences in macular pigment density and distribution. Invest Ophthalmol Vis Sci. 2007 Aug;48(8):3783-7. doi: 10.1167/iovs.06-1218. PMID 17652752
- [Background] Isaacs B, Akhtar AJ. The set test: a rapid test of mental function in old people. Age Ageing. 1972 Nov;1(4):222-6. doi: 10.1093/ageing/1.4.222. No abstract available. PMID 4669878
- [Background] Amieva H, Le Goff M, Millet X, Orgogozo JM, Peres K, Barberger-Gateau P, Jacqmin-Gadda H, Dartigues JF. Prodromal Alzheimer's disease: successive emergence of the clinical symptoms. Ann Neurol. 2008 Nov;64(5):492-8. doi: 10.1002/ana.21509. PMID 19067364
- [Background] Samieri C, Feart C, Proust-Lima C, Peuchant E, Dartigues JF, Amieva H, Barberger-Gateau P. omega-3 fatty acids and cognitive decline: modulation by ApoEepsilon4 allele and depression. Neurobiol Aging. 2011 Dec;32(12):2317.e13-22. doi: 10.1016/j.neurobiolaging.2010.03.020. Epub 2010 Jun 8. PMID 20570406
- [Derived] Korobelnik JF, Rougier MB, Delyfer MN, Bron A, Merle BMJ, Savel H, Chene G, Delcourt C, Creuzot-Garcher C. Effect of Dietary Supplementation With Lutein, Zeaxanthin, and omega-3 on Macular Pigment: A Randomized Clinical Trial. JAMA Ophthalmol. 2017 Nov 1;135(11):1259-1266. doi: 10.1001/jamaophthalmol.2017.3398. PMID 28973076